CLINICAL TRIAL: NCT05516693
Title: Characterization of Chewing and Swallowing and Verification of the Effectiveness of Orofacial Motricity Stimulation in Severe Obese Pre and Post Bariatric Surgery: a Randomized Controlled Clinical Trial.
Brief Title: Chewing, Swallowing and Orofacial Motricity in Severe Obese
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário de Anapolis (Other)
Collaborators: Centro Universitário Fundação Assis Gurgacz (Unknown)
Responsible Party: Principal Investigator, Luis Vicente Franco de Oliveira, Coordinator, Centro Universitário de Anapolis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniEv005/22
Record Dates: First submitted 2022-05-02; First posted 2022-08-25 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Mastication Disorder; Swallowing Disorder; Orofacial Dyskinesia
Keywords: Mastication Disorder; Swallowing Disorder; Orofacial Dyskinesia
MeSH Terms: conditions — Deglutition Disorders; Dyskinesias

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled clinical trial with two intervention arms, involving severely obese adult patients of both sexes referred for bariatric surgery.
Who Masked: Outcomes Assessor
Masking Description: The Outcomes Advisor will be blind to the analysis of the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (MOG) (Experimental): Patients in the experimental group (MOG) will undergo a myofunctional training protocol.
  Interventions: Other: Myofacial muscle training protocol.
- Control group (COG) (No Intervention): Patients in the control group (COG) will not undergo any intervention, being only evaluated at the beginning and at the end of the protocol.

INTERVENTIONS:
Other: Myofacial muscle training protocol. — Muscle training for orofacial motricity stimulation
  Arms: Intervention group (MOG)

SUMMARY:
Background: Obesity is considered an epidemic disease of great repercussion on the world and its prevalence has increased in recent decades. The treatment of obesity aims to improve health and quality of life, by reducing body weight. The clinical approach to obesity is routinely the first line of treatment. Clinical treatment usually involves a combination of restriction of caloric intake, modification of behavior and habits, regular practice of physical activity and pharmacotherapy. Clinical treatment of obesity leads to considerable weight loss, but often not sustained in most patients. This long-term sustained weight loss is an attribute of bariatric surgery, since severe obesity remains largely refractory to dietary and drug therapy. Changes in lifestyle that occur in severely obese patients undergoing bariatric surgery, especially in terms of food, lead to the need for the contribution of speech therapy to adapt to the new way of ingesting food. Objectives: to analyze the stomatognathic functions of mastication and swallowing and to verify the effectiveness of orofacial motricity stimulation in adults, severely obese before and after bariatric surgery. Methods: This is a randomized, controlled clinical trial involving severely obese adult patients of both sexes referred for bariatric surgery. This study was approved by the Research Ethics Committee of the Centro Universitário Fundação Assis Gurgacz (FAG) in the city of Cascavel (PR), Brazil, protocol number CEP FAG no. 4,169,295. Patients will be consecutively recruited from the Bariatric Surgery Department of Hospital São Lucas (FAG) and referred to the Speech Therapy Clinic according to the eligibility criteria of the research protocol. After the initial assessment, patients will be randomly assigned to an intervention group (MOG) and a control group (COG). The COG and MOG groups will be evaluated before and after bariatric surgery. Only the GMO will be submitted to the speech therapy training program before bariatric surgery. The myofunctional characteristics will be evaluated through the Orofacial Myofunctional Assessment protocol with Scores (AMIOFE). The AMIOFE protocol was designed according to the assessment models that reflect the physical characteristics and orofacial behaviors of individuals. In this way, the components and functions of the stomatognathic system will be evaluated in terms of appearance/posture, mobility and swallowing functions - liquid and solid - chewing and breathing.

DETAILED DESCRIPTION:
Obesity is considered an epidemic disease of great repercussion on the world stage and its prevalence has increased in recent decades. It is considered that around 1.9 billion adults worldwide are overweight, of which 600 million are obese. The treatment of obesity aims to improve health and quality of life, by reducing body weight, enough to eliminate or reduce comorbidities and promote psychological well-being. The clinical approach to obesity is routinely the first line of treatment prescribed by medical staff. Clinical treatment usually involves a combination of restriction of caloric intake, modification of behavior and habits, regular practice of physical activity, and pharmacotherapy. Clinical treatment of obesity leads to considerable weight loss but is often not sustained in most patients. This long-term sustained weight loss is an attribute of bariatric surgery since severe obesity remains largely refractory to dietary and drug therapy. Changes in lifestyle that occur in severely obese patients undergoing bariatric surgery, especially in terms of food, lead to the need for the contribution of speech therapy, always aiming at a better quality of life for these individuals. These patients will need to adapt to the new way of ingesting food, paying attention to the particularities of masticatory mechanics. The main objective of this study is to analyze the stomatognathic functions of mastication and swallowing and to verify the effectiveness of orofacial motricity stimulation in adults, severely obese before and after bariatric surgery. As specific objectives, it is intended to characterize the masticatory profile after the oral myofunctional intervention, verify the swallowing function for liquids and solids, measure the quality of life and verify a possible correlation between the variables analyzed before and after bariatric surgery in patients with severe obesity. The hypothesis of this study is based on the masticatory and swallowing profile in severely obese patients before and after bariatric surgery, which will present significant differences in muscle mobility while maintaining functionality without major changes.

This is a randomized, controlled clinical trial involving severely obese adult patients of both sexes referred for bariatric surgery. This study was approved by the Research Ethics Committee of the Centro Universitário Fundação Assis Gurgacz in the city of Cascavel (PR), Brazil, protocol number CEP FAG no. 4,169,295. Patients will be consecutively recruited from the Bariatric Surgery Department of Hospital São Lucas, linked to the Fundação Assis Gurgacz University Center (FAG), and referred to the institution's Speech Therapy Clinic according to the eligibility criteria of the research protocol.

The inclusion criteria will be patients with severe obesity, candidate for bariatric surgery, and participant of the Unified Health System (SUS) of the Department of Bariatric Surgery of Hospital São Lucas. Both sexes, aged over 18 years, agreed to participate in the study and signed the Free and Informed Consent Form (FICT). The exclusion criteria will be patients with significant dental alterations, without the use of dental prostheses; diagnosed temporomandibular joint disorders; patients with clinical and/or mental instability; cerebrovascular disease; any type of active cancer and patients with psychopathies and/or psychiatric illness.

After the initial assessment, patients will be randomly assigned to an intervention group (GMO) and a control group (GCO). The numbers for randomization will be created from a random table in the Speech-Language Pathology and Audiology Laboratory-FAG. In this place, a sequence of sealed, opaque, and serial numbered envelopes will be created, thus ensuring secrecy. Each envelope will contain a card, with the inscription of which group the patient should participate. After randomization of patients, the GMO intervention group will use oral myofunctional therapy as clinically indicated, for 60 days before bariatric surgery.

The GCO and GMO groups will be evaluated before and after bariatric surgery. Only the GMO will be submitted to the speech therapy training program before bariatric surgery. After bariatric surgery, all subjects will be reassessed. The clinical evaluation of oral motricity will be performed through palpation of the masseter and temporal muscles. The myofunctional characteristics will be evaluated through visual inspection, using the Orofacial Myofunctional Assessment protocol with Scores (AMIOFE). The AMIOFE protocol was designed according to the assessment models, with the addition of numerical scales that reflect the physical characteristics and orofacial behaviors of individuals. In this way, the components and functions of the stomatognathic system will be evaluated in terms of appearance/posture, mobility, and swallowing functions - liquid and solid - chewing and breathing.

Exercises involving the oral structures, lips, tongue, and orofacial muscles will be defined for each patient, according to the AMIOFE Protocol, and according to the functionality and needs of each patient. The myofunctional characteristics will be evaluated by a speech therapist, researcher of the study, through visual inspection.

The clinical evaluation of oral motricity will be performed through palpation of the masseter and temporal muscles. Following the standardized protocol for collection has proved to be an efficient method of analyzing the muscles of the stomatognathic system, showing good diagnostic reproducibility, with consistent results. For the analysis of the chewing function, the patients will be instructed to chew a cracker of water and salt, in a usual way, being observed the crushing, the presence of associated body movements, if there is food leakage if the crushing is bilateral, alternating or one-sided.

For the behavior of the tongue, it will be observed if it is contained in the oral cavity or if there is light or excess interposition between the dental arches due to adaptation or dysfunction. Swallowing efficiency, considered in this case as the ability to push the bolus from the oral cavity to the oropharynx, will be evaluated for solid and liquid swallowing. The order to start chewing will be given by the examiner and will start the evaluation process when the mouth is opened to start the chewing process and will be stopped when the cookie is completely swallowed. For swallowing, 8 ml of water will be collected in a glass and the evaluated will be instructed to swallow the liquid when requested. The speech therapist will perform cervical auscultation during swallowing. The order to swallow will be given by the examiner, the evaluated will swallow at once. The process will be carried out within the estimated time of 30 seconds.

In this study, the AMIOFE protocol will be used for the assessment of oral motricity and the WHOQOL Bref quality of life questionnaire considering the physical, psychological, social relationships, and environment domains.

The clinical evaluation will be carried out by doctors (clinicians and surgeons) belonging to the hospital outpatient environment, always by the same team of the services involved. This evaluation will consist of clinical anamnesis, verification of vital signs heart rate, respiratory rate, peripheral arterial pressures (BP), body weight, height, body mass index (BMI) calculated using the weight/height formula2, verification of waist circumferences, hip and neck.

The data obtained will be coded and entered into a database created in Excel and SPSS 23.1 programs and will be analyzed both quantitatively and qualitatively, being presented as mean ± standard deviation, median, and quartile intervals, when applicable. To compare continuous variables before and after the use of myofunctional therapy paired Student's t-test or Wilcoxon test will be used, as appropriate. Comparisons between groups will be performed using Student's t-test or Mann-Whitney U test, according to their distribution. All tests will be two-tailed and p-values less than 0.05 assumed to represent statistical significance. Repeated measurements will be analyzed using analysis of variance (ANOVA) and correlations will be performed using Pearson's method. All analyzes will be performed using SPSS software version 23.1. By monitoring the proposed schedule, we will be developing and evaluating the proposed research activities to maintain quality control.

ELIGIBILITY:
Inclusion criteria:

* severe obesity, candidates for bariatric surgery, participants in the Bariatric Surgery program at Hospital São Lucas;
* both genders;
* over 18 years of age;
* agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* significant dental changes and/or use of dental prostheses
* temporomandibular joint alterations
* clinical and/or mental instability
* sequelae of cerebrovascular disease
* any active cancer;
* pregnancy;
* psychopathies and/or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Masticatory and swallowing profile | 1 year
  Orofacial Myofunctional Assessment Protocol with scores ranging from 0 to 4, the closer to four, the higher the normality index.

CONTACTS AND LOCATIONS:
Overall Officials: Luis VF Oliveira, PhD, Study Chair — University Center of Anápolis
Locations (1):
- Centro Universitário de Anápolis - UniEVANGÉLICA, Anápolis, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After the end of the study, the data will be available to other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the end of the study.
Access Criteria: As per request.
URL: https://www.fag.edu.br/fonoaudiologia